CLINICAL TRIAL: NCT01665911
Title: An in Situ Study on the Impact of Fluoride Dose and Concentration in Milk on Its Anti-caries Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frank Lippert (Other)
Collaborators: The Borrow Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Frank Lippert, Assistant Research Professor, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 12-I-086
Record Dates: First submitted 2012-08-07; First posted 2012-08-16 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Caries
Keywords: Caries
MeSH Terms: interventions — Sodium Fluoride; Milk

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Other): non-fluoridated milk, 200 ml 1.5 mg sodium fluoride in 100 ml milk, 1.5 mg sodium fluoride in 200 ml milk, 3 mg sodium fluoride in 100 ml milk, 3 mg sodium fluoride in 200 ml milk
  Interventions: Drug: 1.5 mg Sodium Fluoride in 100 ml milk; Drug: 1.5 mg sodium fluoride in 200 ml milk; Drug: 3 mg sodium fluoride in 100 ml milk; Drug: 3 mg sodium fluoride in 200 ml milk; Other: Non-fluoridated milk, 200 ml
- Arm 2 (Other): non-fluoridated milk, 200 ml 1.5 mg sodium fluoride in 100 ml milk, 1.5 mg sodium fluoride in 200 ml milk, 3 mg sodium fluoride in 100 ml milk, 3 mg sodium fluoride in 200 ml milk
  Interventions: Drug: 1.5 mg Sodium Fluoride in 100 ml milk; Drug: 1.5 mg sodium fluoride in 200 ml milk; Drug: 3 mg sodium fluoride in 100 ml milk; Drug: 3 mg sodium fluoride in 200 ml milk; Other: Non-fluoridated milk, 200 ml
- Arm 3 (Other): non-fluoridated milk, 200 ml 1.5 mg sodium fluoride in 100 ml milk, 1.5 mg sodium fluoride in 200 ml milk, 3 mg sodium fluoride in 100 ml milk, 3 mg sodium fluoride in 200 ml milk
  Interventions: Drug: 1.5 mg Sodium Fluoride in 100 ml milk; Drug: 1.5 mg sodium fluoride in 200 ml milk; Drug: 3 mg sodium fluoride in 100 ml milk; Drug: 3 mg sodium fluoride in 200 ml milk; Other: Non-fluoridated milk, 200 ml
- Arm 4 (Other): non-fluoridated milk, 200 ml 1.5 mg sodium fluoride in 100 ml milk, 1.5 mg sodium fluoride in 200 ml milk, 3 mg sodium fluoride in 100 ml milk, 3 mg sodium fluoride in 200 ml milk
  Interventions: Drug: 1.5 mg Sodium Fluoride in 100 ml milk; Drug: 1.5 mg sodium fluoride in 200 ml milk; Drug: 3 mg sodium fluoride in 100 ml milk; Drug: 3 mg sodium fluoride in 200 ml milk; Other: Non-fluoridated milk, 200 ml
- Arm 5 (Active Comparator): non-fluoridated milk, 200 ml 1.5 mg sodium fluoride in 100 ml milk, 1.5 mg sodium fluoride in 200 ml milk, 3 mg sodium fluoride in 100 ml milk, 3 mg sodium fluoride in 200 ml milk
  Interventions: Drug: 1.5 mg Sodium Fluoride in 100 ml milk; Drug: 1.5 mg sodium fluoride in 200 ml milk; Drug: 3 mg sodium fluoride in 100 ml milk; Drug: 3 mg sodium fluoride in 200 ml milk; Other: Non-fluoridated milk, 200 ml

INTERVENTIONS:
Drug: 1.5 mg Sodium Fluoride in 100 ml milk — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Other Names: sodium fluoride (PCCA Sodium Fluoride USP 51927-1038-00); Kroger Nonfat Dry Milk reconstituted with fluoride-free milk
Drug: 1.5 mg sodium fluoride in 200 ml milk — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Other Names: sodium fluoride (PCCA Sodium Fluoride USP 51927-1038-00); Kroger Nonfat Dry Milk reconstituted with fluoride-free milk
Drug: 3 mg sodium fluoride in 100 ml milk — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Other Names: sodium fluoride (PCCA Sodium Fluoride USP 51927-1038-00); Kroger Nonfat Dry Milk reconstituted with fluoride-free milk
Drug: 3 mg sodium fluoride in 200 ml milk — Each subject will use this product during one of the five treatment periods in the crossover study design
  Other Names: sodium fluoride (PCCA Sodium Fluoride USP 51927-1038-00); Kroger Nonfat Dry Milk reconstituted with fluoride-free milk
Other: Non-fluoridated milk, 200 ml — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Other Names: Kroger Nonfat Dry Milk

SUMMARY:
The study will be randomized, investigator-blind, observer-blind, laboratory analyst-blind and will utilize a 5-way cross-over study design with a primary objective to determine if a higher dose of fluoride in milk will provide a greater caries preventive effect. Secondary objectives are to determine in a higher concentration of fluoride in milk will provide a greater caries preventive effect and if the caries preventive effect of fluoridated milk follows a dose-response pattern.

DETAILED DESCRIPTION:
The evidence of milk fluoridation as a public health measure in caries prevention has been demonstrated in many clinical studies. While these data are encouraging, the main focus now should be on the optimization of milk fluoride programs. This protocol will concentrate on the parameters of fluoride dose and concentration utilizing an in situ model, the intra-oral caries test or model (ICT). The ICT is an established model which features the use of gauze-covered specimens to facilitate plaque growth and to simulate a caries-prone/plaque stagnation area. After subject has been consented and enrolled in the study per the inclusion/exclusion criteria, two to three days following a dental cleaning, two partially demineralized specimens will be placed in the buccal flange area of the subject's mandibular partial denture. During each of the five, three-week test periods, subjects will drink their assigned milk test product once per day for either five (100 ml milk) or ten (200 ml milk) timed minutes, wearing their mandibular partial dentures 24 hours a day during the test period. Fluoride free toothpaste will be used two to three days before and continuously during each treatment period. After each three-week test period, the two partially demineralized specimens will be removed from the subject's partial denture and analyzed using the surface microhardness test. Mineral content change (as percentage of surface microhardness recovery) in these artificially induced incipient enamel lesions will be the primary outcome variable. Each subject (n = 28) will serve as his or her own control.

ELIGIBILITY:
Inclusion Criteria:

* sign an informed consent, authorization for the release of health information for research and provide medical history information, including medications, prior to their participation;
* be between 18 and 80 years old and in general good health;
* willingness to use a reliable form of contraception or abstaining during the course of the study (females of child-bearing potential only)
* wear a removable mandibular partial denture with sufficient room in one posterior buccal flange area to accommodate two enamel specimens (required dimensions 12×7 mm);
* be willing and capable of wearing their removable mandibular partial dentures 24 hours a day for a total of five, three-week test periods;
* be in good dental health with no active caries or periodontal disease;
* agree to comply with all subjects' responsibilities as stated in the protocol (e.g. use of study products, attendance at appointments, etc.);
* have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 ml/min; gum base stimulated whole saliva flow rate ≥ 0.8 ml/min).
* Be able to tolerate the taste and room temperature of the mixed milk product as demonstrated by drinking the milk at screening

Exclusion Criteria:

be pregnant, intending to become pregnant during the study period or breast feeding. A urine pregnancy test will be required at screening, the start of each treatment visit and the last study visit for all subjects of child-bearing potential to confirm the subject is not pregnant.

* have any medical condition that could be expected to interfere with the subject's safety during the study period;
* demonstrate an inability to comply with study procedures;
* have factors which could contraindicate their participation, such as any condition requiring the need for antibiotic premedication prior to a dental treatment, a condition requiring the need for long-term antibiotic use, blood thinning medications that prohibit the safe conduct of a dental cleaning* or previous use of the weight loss medications Fen Phen® or Redux®. (*Note: Subjects who are taking blood thinners in which written verification is obtained from their physician indicating their PT/INR levels (anti-coagulation blood levels) are at an acceptable level to avoid serious complications, such as bleeding during dental cleanings, may be accepted into the study at the discretion of the Investigator.)
* be currently taking or have ever taken a bisphosphonate drug (i.e. Fosamax®, Actonel®, Boniva®, Reclast®, or Zometa®) for treatment of osteoporosis.
* be lactose intolerant or have known allergy or intolerance to milk or milk products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lippert, PhD, Principal Investigator — Indiana University; Domenick Zero, DDS, MS, Principal Investigator — Indiana University
Locations (1):
- Oral Health Research Institute, Indiana University School of Dentistry, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Lippert F, Martinez-Mier EA, Zero DT. An in situ caries study on the interplay between fluoride dose and concentration in milk. J Dent. 2014 Jul;42(7):883-90. doi: 10.1016/j.jdent.2014.01.010. Epub 2014 Feb 7. PMID 24513113

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Each subject will use each of these products during each of the five treatment periods in the crossover study design. There were five interventions as follows:
  1. . 1.5 mg Sodium Fluoride in 100 ml milk: .
  2. 1.5 mg Sodium Fluoride in 200 ml milk
  3. 3.0 mg Sodium Fluoride in 100 ml milk
  4. 3.0 mg Sodium Fluoride in 200 ml milk
  5. 0 mg fluoride in 200 ml milk
Period: Overall Study
Arm/Group | All Participants
Started | 28
0 mg Fluoride in 200 ml Milk | 22
1.5 mg Sodium Fluoride in 100 ml Milk | 23
1.5 mg Sodium Fluoride in 200 ml Milk | 25
3.0 mg Sodium Fluoride in 100 ml Milk | 22
3.0 mg Sodium Fluoride in 200 ml Milk | 22
Completed | 22
Not Completed | 6
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: 1. 1.5 mg Sodium Fluoride in 100 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design.
  2. 1.5 mg sodium fluoride in 200 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design.
  3. 3 mg sodium fluoride in 100 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design.
  4. 3 mg sodium fluoride in 200 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design
  5. Non-fluoridated milk, 200 ml: Each subject will use this product during one of the five treatment periods in the crossover study design
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: % Surface Microhardness (SMH) Recovery Score Per Each of Five Arms
Description: * surface microhardness recovery is a measure of caries lesion remineralization and is calculated using the following equation:
  * SMHr=(D1-R)/(D1-B)×100 B = indentation length of sound enamel specimen at baseline D1 = indentation length after first in vitro demineralization R = indentation length after intra-oral exposure (rehardening).
Time Frame: Three Weeks per each of five arms
Measure: Least Squares Mean (Standard Error); unit: percent
Groups:
- All Participants: 1.5 mg sodium fluoride in 100 ml milk 1.5 mg sodium fluoride in 200 ml milk 3 mg sodium fluoride in 100 ml milk 3 mg sodium fluoride in 200 ml milk non-fluoridated milk, 200 ml
  Each of the subjects used all of the five inverventions listed above during this 5-period cross over study. Each subject had their own specific sequence of use.
Arm/Group | All Participants
Number analyzed (Participants) | 22
percent
  0 mg fluoride in 200 ml milk | 20 (2)
  1.5 mg fluoride in 100 ml milk | 24 (2)
  1.5 mg fluoride in 200 ml milk | 22.5 (1.9)
  3.0 mg fluoride in 100 ml milk | 26.7 (2)
  3.0 mg fluoride in 200 ml milk | 25.4 (2)
Statistical Analysis 1: Comparison: All Participants; Based on prior studies using a variety of products in this model, the within-product standard deviation of %SMH recovery is estimated to be 13% and the correlation between products is expected to be approximately 0.5. With a sample size of 28 subjects in a 5-way crossover study, the study will have 80% power to detect a %SMH recovery difference of 8.6%, assuming two-sided tests each conducted at a 5% significance level; Test type: Superiority or Other; p = 0.0490, ANOVA — Non-fluoridated milk, 200 ml vs. 1.5 mg Sodium Fluoride in 100 ml milk
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; p = 0.19, ANOVA — Non-fluoridated milk, 200 ml vs. 1.5 mg sodium fluoride in 200 ml milk
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority or Other; p = 0.0017, ANOVA — Non-fluoridated milk, 200 ml vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 4: Comparison: All Participants; Test type: Superiority or Other; p = 0.0092, ANOVA — Non-fluoridated milk, 200 ml vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 5: Comparison: All Participants; Test type: Superiority or Other; p = 0.45, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 1.5 mg sodium fluoride in 200 ml milk
Statistical Analysis 6: Comparison: All Participants; Test type: Superiority or Other; p = 0.18, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 7: Comparison: All Participants; Test type: Superiority or Other; p = 0.47, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 8: Comparison: All Participants; Test type: Superiority or Other; p = 0.0423, ANOVA — 1.5 mg sodium fluoride in 200 ml milk vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 9: Comparison: All Participants; Test type: Superiority or Other; p = 0.15, ANOVA — 1.5 mg sodium fluoride in 200 ml milk vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 10: Comparison: All Participants; Test type: Superiority or Other; p = 0.54, ANOVA — 3 mg sodium fluoride in 100 ml milk vs. 3 mg sodium fluoride in 200 ml milk

2. Secondary Outcome: % Acid Resistance Score Per Each of Five Arms
Description: % Acid Resistance is a measure of acid resistance of the remineralized caries lesion which is calculated as (D1-D2)/(D1-B)*100%, where B is the indentation length of sound enamel specimen at baseline, D1 is an indentation length after first in vitro demineralization, D2 is an indentation length after second in vitro demineralization.
Time Frame: Three Weeks per each of five arms
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | All Participants
Number analyzed (Participants) | 22
percent
  0 mg fluoride in 200 ml milk | -3.4 (2.0)
  1.5 mg fluoride in 100 ml milk | 2.6 (2.0)
  1.5 mg fluoride in 200 ml milk | -0.2 (1.9)
  3.0 mg fluoride in 100 ml milk | 5.4 (2.0)
  3.0 mg fluoride in 200 ml milk | 6.0 (2.0)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.24, ANOVA — Non-fluoridated milk, 200 ml vs. 1.5 mg Sodium Fluoride in 100 ml milk
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; p = 0.17, ANOVA — Non-fluoridated milk, 200 ml vs. 1.5 mg sodium fluoride in 200 ml milk
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority or Other; p = 0.0008, ANOVA — Non-fluoridated milk, 200 ml vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 4: Comparison: All Participants; Test type: Superiority or Other; p = 0.0003, ANOVA — Non-fluoridated milk, 200 ml vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 5: Comparison: All Participants; Test type: Superiority or Other; p = 0.24, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 1.5 mg Sodium Fluoride in 200 ml milk
Statistical Analysis 6: Comparison: All Participants; Test type: Superiority or Other; p = 0.26, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 7: Comparison: All Participants; Test type: Superiority or Other; p = 0.18, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 8: Comparison: All Participants; Test type: Superiority or Other; p = 0.0269, ANOVA — 1.5 mg sodium fluoride in 200 ml milk vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 9: Comparison: All Participants; Test type: Superiority or Other; p = 0.0142, ANOVA — 1.5 mg sodium fluoride in 200 ml milk vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 10: Comparison: All Participants; Test type: Superiority or Other; p = 0.81, ANOVA — 3 mg sodium fluoride in 100 ml milk vs. 3 mg sodium fluoride in 200 ml milk

3. Secondary Outcome: Enamel Fluoride Uptake Per Each of Five Arms
Description: Enamel fluoride uptake is a measure of fluoridation of a caries lesion
Time Frame: Three Weeks per each of five arms
Measure: Least Squares Mean (Standard Error); unit: microgram fluoride per square cm
Arm/Group | All Participants
Number analyzed (Participants) | 22
microgram fluoride per square cm
  0 mg fluoride in 200 ml milk | 1.2 (0.18)
  1.5 mg fluoride in 100 ml milk | 2.4 (0.17)
  1.5 mg fluoride in 200 ml milk | 2.12 (0.17)
  3.0 mg fluoride in 100 ml milk | 3.09 (0.18)
  3.0 mg fluoride in 200 ml milk | 2.67 (0.18)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.0000, ANOVA — Non-fluoridated milk, 200 ml vs. 1.5 mg Sodium Fluoride in 100 ml milk
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; p = 0.0000, ANOVA — Non-fluoridated milk, 200 ml vs. 1.5 mg sodium fluoride in 200 ml milk
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority or Other; p = 0.0000, ANOVA — Non-fluoridated milk, 200 ml vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 4: Comparison: All Participants; Test type: Superiority or Other; p = 0.0000, ANOVA — Non-fluoridated milk, 200 ml vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 5: Comparison: All Participants; Test type: Superiority or Other; p = 0.14, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 1.5 mg Sodium Fluoride in 200 ml milk
Statistical Analysis 6: Comparison: All Participants; Test type: Superiority or Other; p = 0.0012, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 7: Comparison: All Participants; Test type: Superiority or Other; p = 0.19, ANOVA — 1.5 mg Sodium Fluoride in 100 ml milk vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 8: Comparison: All Participants; Test type: Superiority or Other; p = 0.0000, ANOVA — 1.5 mg sodium fluoride in 200 ml milk vs. 3 mg sodium fluoride in 100 ml milk
Statistical Analysis 9: Comparison: All Participants; Test type: Superiority or Other; p = 0.0075, ANOVA — 1.5 mg sodium fluoride in 200 ml milk vs. 3 mg sodium fluoride in 200 ml milk
Statistical Analysis 10: Comparison: All Participants; Test type: Superiority or Other; p = 0.0444, ANOVA — 3 mg sodium fluoride in 100 ml milk vs. 3 mg sodium fluoride in 200 ml milk

ADVERSE EVENTS:
Time Frame: Six months
Groups:
- Arm/Group All Participants: 1.5 mg sodium fluoride in 100 ml milk 1.5 mg sodium fluoride in 200 ml milk 3 mg sodium fluoride in 100 ml milk 3 mg sodium fluoride in 200 ml milk non-fluoridated milk, 200 ml
  1.5 mg Sodium Fluoride in 100 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design.
  1.5 mg sodium fluoride in 200 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design.
  3 mg sodium fluoride in 100 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design.
  3 mg sodium fluoride in 200 ml milk: Each subject will use this product during one of the five treatment periods in the crossover study design
  Non-fluoridated milk, 200 ml: Each subject will use this product during one of the five treatment periods in the crossover study design.
Arm/Group | Arm/Group All Participants
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No